CLINICAL TRIAL: NCT05309304
Title: Pharmacokinetic Study of Cefazolin 3 g/150 mL in Subjects Weighing Greater Than or Equal to 120 kg Versus Cefazolin 2 g/100 mL in Subjects Weighing Less Than 120 kg
Brief Title: Cefazolin PK Study 3g vs 2g
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Baxter Healthcare Corporation (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: BXU567633
Record Dates: First submitted 2022-03-25; First posted 2022-04-04 (Actual); Last update posted 2022-10-12 (Actual); Status verified 2022-10

CONDITIONS: Healthy
MeSH Terms: interventions — Cefazolin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- 3 g cefazolin (Experimental): Healthy adult subjects weighing ≥120 kg. (g=grams)
  Interventions: Drug: Cefazolin
- 2 g cefazolin (Active Comparator): Healthy adult subjects weighing <120 kg. (g=grams)
  Interventions: Drug: Cefazolin

INTERVENTIONS:
Drug: Cefazolin — Cefazolin Injection - 2 g/100 mL or 3 g/150 mL

SUMMARY:
Study is to characterize the safety and tolerability of cefazolin after a single IV administration in healthy subjects in a 3 g/150 mL presentation to meet the increasing clinical need for the indication of perioperative prophylaxis in this patient population weighing greater than or equal to (≥) 120 kg.

ELIGIBILITY:
Inclusion Criteria:

* Subject provides informed consent (approved by an Institutional Review Board [IRB]) before any study specific evaluation is performed.
* Subject is between the ages of 18 and 55 years (both inclusive).
* A female subject is eligible to participate if she is not pregnant, breastfeeding, and not planning to become pregnant at Screening and upon Admission to the clinic.
* Subject must agree to use an adequate method of contraception

  * For male subjects: Subjects willing to follow approved birth control methods (a double barrier method) from signed ICF to Follow up call as judged by the Investigator(s), such as condom with spermicide, condom with diaphragm, or abstinence. Subjects should also not donate sperm during this time.
  * For female subjects: Female subjects of childbearing potential, defined as a woman ≤ 55 years of age who has not had a partial or full hysterectomy or oophorectomy, must have a negative serum beta-human chorionic gonadotropin (β-hCG) pregnancy test at Screening and Admission. Subjects of childbearing potential must use a medically acceptable means of contraception from signed ICF to Follow up call. Subjects should also not participate in egg donation during this time.
* Subject must, in the opinion of the Investigator, be in good health based upon medical history, physical examination (including vital signs) and clinical laboratory tests assessed at the time of Screening.
* Subject is a nonsmoker or has quit smoking at least 6 months before the dose of study drug.

Exclusion Criteria:

* Subject has a known history of hypersensitivity to cefazolin, any of its components, or any beta lactam antibiotic.
* Subject has active or recurring clinically significant renal, hepatic, skin, head, ears, eyes, nose, throat, respiratory, cardiovascular, gastrointestinal, endocrine/metabolic, genitourinary, neurologic, hematologic, musculoskeletal, immunologic, allergic, psychological/psychiatric, or other disease requiring medical treatment.
* Subject has an active malignancy of any type other than nonmelanomatous skin malignancies.
* Subject has any history of alcohol abuse or drug addiction.
* Subject has a positive test result for drugs of abuse (opiates, methadone, cocaine, amphetamines, cannabinoids, barbiturates, benzodiazepines, tricyclic antidepressants, oxycodone), cotinine, or alcohol.
* Subject has any history of relevant drug and/or food allergies as judged by the Investigator.
* Subjects who have received any IMP in a clinical research study within 5 halflives or within 30 days prior to first dose. However, in no event, shall the time between last receipt of IMP and first dose be less than 30 days.
* Subject has received probenecid within 4 weeks before dosing, or any other overthe-counter medication (including vitamins, herbal supplements, or dietary supplements) within 2 weeks before dosing.
* Subject has donated or lost 550 mL or more of blood (including plasmapheresis) within 60 days before the first dose of study drug.
* Subject has a positive test result for human immunodeficiency virus (HIV; 1 or 2) antibody, hepatitis B surface antigen, or hepatitis C virus antibody.
* Subject has any clinically significant illness within 5 days before the first dose of study drug as judged by the Investigator.
* Subject is a member of the professional or ancillary personnel involved in the study.
* Subject is deemed not suitable for entry into the study in the opinion of the Investigator.
* Failed facility's COVID-19 screening questions or tested positive for COVID-19 in a polymerase chain reaction (PCR) test on Study Day.

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 24 (Actual)
Dates: Start 2022-02-14 (Actual); Primary Completion 2022-08-30 (Actual); Study Completion 2022-08-30 (Actual)

PRIMARY OUTCOMES:
Area under the curve (AUC) | Day 1 (15 minutes prior to dosing as a baseline measurement and at 2, 10, 20, 30, 45, 60, 90, 120, 150, 180, 240, 300,360, 420, and 480 minutes post-dosing)
  Cefazolin in plasma.
Maximum concentration (Cmax) | Day 1 (15 minutes prior to dosing as a baseline measurement and at 2, 10, 20, 30, 45, 60, 90, 120, 150, 180, 240, 300,360, 420, and 480 minutes post-dosing)
  Cefazolin in plasma
Number of subjects with TEAEs | Day 1 to Day 10
  Treatment Emergent Adverse Events (TEAEs)
Number of subjects with Non-serious TEAEs | Day 1 to Day 10
Number of subjects with Serious TEAEs | Day 1 to Day 10
Number of subjects with TEAEs related to study treatment | Day 1 to Day 10
Number of subjects with Serious TEAEs related to study treatment | Day 1 to Day 10
Number of subjects with TEAEs leading to withdrawal | Day 1 to Day 10
Number of subjects with phlebitis at the infusion site | Day 1 to Day 10

CONTACTS AND LOCATIONS:
Locations (1):
- Baxter Investigational Site, Baltimore, Maryland, United States

IPD SHARING:
Plan to Share IPD: Yes
Sharing of Clinical Trial Data: Baxter is committed to sharing clinical trial data with external medical experts and scientific researchers in the interest of advancing public health. As such, Baxter will supply anonymized Individual Patient Datasets (IPD) and supporting documents (synopsis of clinical study reports, protocol and SAP's)
Supporting Information: Study Protocol, SAP, CSR
Time Frame: Upon approval of a legitimate research request.
Access Criteria: Research requests will be reviewed by qualified medical and scientific experts within the company. If Baxter agrees to the release of clinical data for research purposes, the requestor will be required to sign a data sharing agreement (DSA) in order to ensure protection of patient confidentiality and any intellectual property rights of Baxter prior to the release of any data.
URL: https://www.baxter.com/clinical-trial-transparency-and-data-sharing-policy